CLINICAL TRIAL: NCT03135639
Title: Evaluating Transcranial Alternating Current Stimulation (tACS) for Enhancing Creativity
Brief Title: Effects of Alpha tACS
Acronym: PACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-3918
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: tACS; transcranial alternating current stimulation; stimulation; healthy control; alpha oscillations; heart rate variability

STUDY DESIGN:
Intervention Model Description: Each participant will receive sham stimulation or stimulation at their individual alpha frequency (8-12 Hz) during a study visit. The order is randomized (i.e., half of participants will receive sham stimulation during the first stimulation session and half will receive sham stimulation during the second stimulation session).
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, meaning that neither the participant nor the experimenter knows what kind of stimulation the participant is receiving. An unblinded monitor (separate from the staff that interacts with the participant) is responsible for creating the stimulation codes that run each session and for ensuring that these codes worked correctly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Stim followed by Alpha Stim (Experimental): 20 minutes of sham stimulation (sham stim) is followed by a washout period of 20 minutes. 20 minutes of alpha stimulation (alpha stim) is applied next.
  Sham stimulation mimics the physical effects of stimulation, with up to 1 minute of stimulation during the session. Sham stimulation is delivered using the NeuroConn Plus Stimulator Sham.
  Participants will receive 2 mA alternating current stimulation at their individual alpha frequency (8-12 Hz, as determined by the 2 minute resting state EEG) for 20 minutes. Alpha stimulation is delivered using the NeuroConn Plus Stimulator tACS.
  Interventions: Other: NeuroConn Plus Stimulator tACS; Other: NeuroConn Plus Stimulator Sham
- Alpha Stim followed by Sham Stim (Experimental): 20 minutes of alpha stimulation (alpha stim) is followed by a washout period of 20 minutes. 20 minutes of sham stimulation (sham stim) is applied next.
  Participants will receive 2 mA alternating current stimulation at their individual alpha frequency (8-12 Hz, as determined by the 2 minute resting state EEG) for 20 minutes. Alpha stimulation is delivered using the NeuroConn Plus Stimulator tACS.
  Sham stimulation mimics the physical effects of stimulation, with up to 1 minute of stimulation during the session. Sham stimulation is delivered using the NeuroConn Plus Stimulator Sham.
  Interventions: Other: NeuroConn Plus Stimulator tACS; Other: NeuroConn Plus Stimulator Sham

INTERVENTIONS:
Other: NeuroConn Plus Stimulator tACS — Transcranial alternating current stimulation (tACS) is a novel, noninvasive brain stimulation approach in which weak electric currents are applied to the scalp. The electric currents that are applied to the scalp are in a sine-wave pattern.
  Other Names: tACS
Other: NeuroConn Plus Stimulator Sham — For sham stimulation, the participant receives up to 1 minute of tACS stimulation until the stimulation fades. This mimics the same skin sensations that a participant would experience during a tACS session.
  Other Names: Sham tACS

SUMMARY:
**Follow-up Control Study for Creativity Study

Purpose: To investigate the effect of transcranial alternating current stimulation (tACS), a form of noninvasive brain stimulation, in healthy subjects. This experiment is a follow-up to previous tACS studies that used a creativity assessment.

Participants: 35 males and females, at least 18 years of age, without history of major psychiatric/neurological disease or associated medication use, or prior brain surgery/implants.

Procedures (methods): This is a cross-over study design. Participants will undergo a control condition of stimulation (sham or individual alpha, 8-12 Hz, tACS) during electroencephalogram recordings. In addition, pupil diameter, heart rate, and respiration will be measured continuously. This is to study the physiological effects of stimulation.

DETAILED DESCRIPTION:
Participants will report for a study visit. They will review and sign a consent form.

They will first be fitted with two 5x7cm electrodes placed over occipital and parietal cortex (Cz and Oz). They will also be fitted with ECG electrodes as well as a respiration belt. In addition, they will have a 128-channel EEG net placed on their head and pupillometry glasses. Once the participant is fitted with this equipment, they will complete a 2-minute resting state EEG with their eyes closed to determine their individual alpha frequency. Following the individual alpha frequency determination, the participant will fill out an alertness questionnaire, followed by 3 EEG recordings:

1. 5 minute before stimulation recording
2. 20 minute recording during stimulation; either at their individual alpha frequency (between 8 and 12 Hz) or sham stimulation.
3. 5 minute after stimulation recording

Following these three recordings, the participant will have a 20 minute break in which they will read neutral reading material or converse with the study staff, as well as provide a saliva sample to test for brain derived neurotropic factor (BDNF).

After the 20 minute break, the participant will complete the alertness questionnaire, and the three recordings will be completed again. The participant will then be allowed to clean up, be paid, and leave.

------------------------

Clarification for the Experimental Design:

This part of the study is a control condition that will consist of stimulation over occipital and parietal cortex with electrodes over Cz and Oz. Participants will then receive 2mA alternating current stimulation between 8Hz and 12Hz (based on their individual alpha frequency determined by a 2 min eyes closed recording) or sham stimulation for 20 minutes (approximately the duration of the TTCT test) in a resting condition where they will have to focus on a cross hair on a computer screen. EEG will be collected simultaneously during this.

In both conditions, the participants wear a Pupil eye tracking headset, which is commercially available. This allows to monitor eye movements and to obtain physiological relevant measures of the pupil.

To obtain a measure of the heart rate during both conditions, ECG electrodes as part of the EEG acquisition system are placed on the participant's body. Ideally one electrode below the left collarbone and a second below the right chest.

Respiration Effort is measured in both conditions by a SleepSense sleep-lab sensor that is placed with an elastic band over the participants chest and connected to the EEG acquisition system.

Before each session, a questionnaire will be administered to the participant to assess the alertness state.

The entire procedure will be conducted by study personnel with documented training using brain stimulators and EEG.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age

Exclusion Criteria:

* History of major neurological or psychiatric illness, including epilepsy
* Medication use associated with neurological or psychiatric illnesses
* Currently undergoing counseling or psychotherapy treatment for depression, anxiety, eating disorders, PTSD, or other behavior conditions
* First degree relative (parent, sibling, child) with neurological or psychiatric illness (past and present)
* Prior brain surgery
* Head injury
* Any brain devices/implants (including cochlear implants and aneurysm clips)
* Cardiovascular disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram power in alpha band | 5 minute recordings before and after each 20 minute stimulation session during a single study visit.
  Changes in the EEG power in the alpha (8-12 Hz) band before and after stimulation sessions.

SECONDARY OUTCOMES:
Heart Rate Variability | 5 minute recordings before and after each 20 minute stimulation session during a single study visit.
  Change in the ratio between the power in low frequency band and the power in high frequency band. As this outcome variable is a ratio between two items that are measured in microvolt^2, the ratio does not have a unit of measure.
Pupil diameter | 5 minute recordings before and after each 20 minute stimulation session during a single study visit.
  Pupil diameter is associated with arousal. We will look to see what the changes in arousal are before and after stimulation sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available starting from 1 year after publication.
Access Criteria: Data will be available for other publications or other brain stimulation researchers. Sharing is at the discretion of the PI.